CLINICAL TRIAL: NCT07161856
Title: Novel Balloon-Assisted vs Direct Technique in EUS-Guided Gastroenterostomy: A Prospective Multicenter RCT
Brief Title: Novel Balloon-Assisted vs Direct Technique in EUS-Guided Gastroenterostomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHEC2025-284
Record Dates: First submitted 2025-08-14; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Gastric Outlet Obstruction
MeSH Terms: conditions — Gastric Outlet Obstruction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- direct EUS-GE (Active Comparator): The patients will receive EUS-DGE under general anesthesia with endotracheal intubation. Under direct visualization with a gastroscope, a guidewire and/or nasobiliary catheter is passed through the stricture into the jejunum. A mixture of contrast medium and methylene blue is injected to distend the target intestinal loop. An echoendoscope is introduced into the stomach to select the optimal puncture site.
  A 19G or 22G puncture needle is used to puncture the gastric and jejunal walls. Aspiration of fluid confirms the needle tip is in the jejunum, after which the channel is dilated over the guidewire. Using the delivery system of an electrocautery-enhanced fully covered lumen-apposing metal stent (LAMS), the stent is deployed to complete the gastrojejunostomy.
  Interventions: Procedure: direct EUS-GE
- a novel balloon-assisted EUS-GE (Experimental): The patients will receive EUS-NBAGE under general anesthesia with endotracheal intubation. Under direct visualization with a gastroscope, contrast medium is injected to determine the location and length of the stricture. A guidewire is then placed through the stricture into the jejunum, approximately 15 cm distal to the anal side of the stricture. A double-balloon device is inserted over the guidewire. The anal-side balloon is inflated with about 40 mL of air, and under fluoroscopy, the balloon is confirmed to be well inflated. A mixture of contrast medium and methylene blue in a 1:1 dilution is injected into the proximal small intestine through the water injection channel at the proximal end of the catheter. A linear echoendoscope is inserted into the mid-body of the stomach on the greater curvature side to scan the distended small intestine loop. After identifying the distended small intestine loop, a HOT-AXIOS 1.5×1.0cm LAMS is placed under direct visualization.
  Interventions: Procedure: a novel balloon-assisted EUS-GE

INTERVENTIONS:
Procedure: a novel balloon-assisted EUS-GE — The patients will receive EUS-NBAGE under general anesthesia with endotracheal intubation. Under direct visualization with a gastroscope, contrast medium is injected to determine the location and length of the stricture. A guidewire is then placed through the stricture into the jejunum, approximately 15 cm distal to the anal side of the stricture. A double-balloon device is inserted over the guidewire. The anal-side balloon is inflated with about 40 mL of air, and under fluoroscopy, the balloon is confirmed to be well inflated. A mixture of contrast medium and methylene blue in a 1:1 dilution is injected into the proximal small intestine through the water injection channel at the proximal end of the catheter. A linear echoendoscope is inserted into the mid-body of the stomach on the greater curvature side to scan the distended small intestine loop. After identifying the distended small intestine loop, a HOT-AXIOS 1.5×1.0cm LAMS is placed under direct visualization.
  Arms: a novel balloon-assisted EUS-GE
Procedure: direct EUS-GE — The patients will receive EUS-DGE under general anesthesia with endotracheal intubation. Under direct visualization with a gastroscope, a guidewire and/or nasobiliary catheter is passed through the stricture into the jejunum. A mixture of contrast medium and methylene blue is injected to distend the target intestinal loop. An echoendoscope is introduced into the stomach to select the optimal puncture site.
  A 19G or 22G puncture needle is used to puncture the gastric and jejunal walls. Aspiration of fluid confirms the needle tip is in the jejunum, after which the channel is dilated over the guidewire. Using the delivery system of an electrocautery-enhanced fully covered lumen-apposing metal stent (LAMS), the stent is deployed to complete the gastrojejunostomy.
  Arms: direct EUS-GE

SUMMARY:
Gastric outlet obstruction (GOO) refers to mechanical blockage at the pylorus or duodenum, most commonly caused by unresectable malignancies of the stomach, duodenum, or pancreas. At the time of diagnosis, the majority of lesions are no longer amenable to curative resection, and median survival ranges from only 11.3 to 21.3 weeks. Throughout the disease course, patients develop nausea, vomiting, and severe malnutrition, which markedly impair quality of life. Current strategies to relieve obstruction include endoscopic stent placement and surgical gastrojejunostomy; however, each is associated with distinct drawbacks, such as stent occlusion, prolonged operative times, and high complication rates.

Endoscopic ultrasound-guided gastroenterostomy (EUS-GE) is a minimally invasive technique in which a gastric-jejunal anastomosis is created under real-time EUS guidance, bypassing the obstructed segment and establishing a gastrojejunal shortcut. Compared with conventional surgery or endoscopic luminal stenting, EUS-GE offers reduced procedural trauma and lower recurrence rates, providing GOO patients with an additional, less-invasive therapeutic option.

Three main EUS-GE approaches have been described: the direct method, the balloon-assisted method, and the double-balloon-assisted method. The direct method requires large volumes of water instillation, posing hemodynamic risks in patients with cardiovascular or cerebrovascular disease. The double-balloon technique relies on expensive, specialized devices that have not yet been widely adopted. The conventional balloon-assisted method demands needle puncture of a partially inflated balloon, which compromises stability and can displace the target jejunum away from the gastric wall. All three techniques are technically demanding, limiting their broad clinical dissemination.

The investigators therefore designed and previously reported a dedicated single-balloon-assisted device specifically for EUS-GE. This novel system aims to shorten procedure time, reduce intraprocedural water volume, and enhance procedural safety. The present prospective, multicenter, randomized controlled trial was undertaken to validate the clinical efficacy and safety of this new single-balloon-assisted technique compared with the conventional direct water-injection method.

DETAILED DESCRIPTION:
This multicenter, single-blind, RCT is designed to enroll 272 patients across five high-volume tertiary referral centers in China. The study is planned to commence in July 2025 and continue until the final patient completed 12 months of follow-up or passed away. The primary outcome is the operation duration. Secondary outcomes are technical success rate, clinical success rate, intraoperative water injection volume, quality of life assessment, length of hospital stay, and incidence of adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* Age ranges from 18 to 80 years old
* GOO patients caused by all reasons (including benign diseases such as ulcers or malignant tumors)
* Not suitable for or cannot tolerate surgical operations and endoscopic intestinal stent implantation
* There are no absolute contraindications for EUS-GE
* Signed informed consents

Exclusion Criteria:

* Pregnant and lactating women
* Unable or refused to provide informed consents
* Patients with cognitive impairment, aphasia, mental disorders, or other conditions that may affect the patient's cooperation
* Patients with endoscopic contraindications, anesthesia contraindications, digestive tract perforation or abdominal cavity infection
* The tumor invades the duodenum or the upper segment of the jejunum Individuals whom the investigator deems unsuitable for participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
operation duration | Perioperative
  the duration from the moment the surgical instrument enters the body and begins operation until the completion of the gastrojejunostomy and placement of the intraluminal stent

SECONDARY OUTCOMES:
technical success | Perioperative
  successfully pass through the narrow intestinal segment and implant the stent, that is, the LAMS stent fully expands and is confirmed through a combination of endoscopy, ultrasound and fluorescence microscopy

IPD SHARING:
Plan to Share IPD: Yes
Primary and secondary outcome measures could be shared without sharing patient privacy. Interested parties can contact by email
Supporting Information: Study Protocol